CLINICAL TRIAL: NCT02081599
Title: A Phase IV Study of Teneligliptin (MP-513) in Combination With Insulin in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of Teneligliptin (MP-513) in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3000-A15
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneli (Teneligliptin) /Teneli + insulin (Experimental): Teneligliptin for 16 weeks (double-blind period) followed by teneligliptin for an additional 36 weeks (open-label period) in combination with insulin.
  Interventions: Drug: Teneli (Teneligliptin); Drug: Insulin
- Placebo/Teneli (Teneligliptin) + insulin (Placebo Comparator): Placebo for 16 weeks (double-blind period) followed by teneligliptin for an additional 36 weeks (open-label period) in combination with insulin.
  Interventions: Drug: Teneli (Teneligliptin); Drug: Placebo; Drug: Insulin

INTERVENTIONS:
Drug: Teneli (Teneligliptin)
Drug: Placebo
  Arms: Placebo/Teneli (Teneligliptin) + insulin
Drug: Insulin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Teneligliptin in combination with Insulin in patients with type 2 Diabetes for 16 weeks administration and to evaluate the safety and efficacy of Teneligliptin in combination with Insulin with an extension treatment for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has been receiving a stable dose and regimen of insulin over 12 weeks before administration of investigational drug
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 12 weeks before administration of investigational drug
* Patients whose HbA1c is between 7.5% and 10.5%
* Patients who were not administered diabetes therapeutic drugs prohibited for concomitant use within 12 weeks before administration of investigational drug.

Exclusion Criteria:

* Patients with type 1 diabetes, diabetes mellitus caused by pancreas impairment, or secondary diabetes (Cushing disease, acromegaly, etc)
* Patients who are accepting treatments of arrhythmias
* Patients with serious diabetic complications
* Patients who are the excessive alcohol addicts
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are pregnant, lactating, and probably pregnant patients, and patients who can not agree to contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, Professor, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Result] Kadowaki T, Kondo K, Sasaki N, Miyayama K, Yokota S, Terata R, Gouda M. Efficacy and safety of teneligliptin add-on to insulin monotherapy in Japanese patients with type 2 diabetes mellitus: a 16-week, randomized, double-blind, placebo-controlled trial with an open-label period. Expert Opin Pharmacother. 2017 Sep;18(13):1291-1300. doi: 10.1080/14656566.2017.1359259. Epub 2017 Aug 10. PMID 28741385

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Teneli (Teneligliptin) + Insulin: Placebo for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained ) for an additional 36 weeks (open-label period) in combination with insulin.
- Teneli (Teneligliptin) /Teneli + Insulin: Teneligliptin (20 mg once daily) for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained ) for an additional 36 weeks (open-label period) in combination with insulin.
Period: Period 1：Double-blind Period
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Started | 71 | 77
Completed | 63 | 75
Not Completed | 8 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — stopping criteria | 1 | 0
Period: Period 2：Open-label Period
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Started | 63 | 75
Completed | 57 | 71
Not Completed | 6 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 2 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin | Total
Number analyzed (Participants) | 71 | 77 | 148
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 49 | 46 | 95
  >=65 years | 22 | 31 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 53 | 59 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 16. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate.
Time Frame: at Week 0 and Week 16
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization. Analysis based on last observation carried forward, where the last post baseline double-blind observed value was carried forward and used for Week 16 where data was missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Number analyzed (Participants) | 71 | 77
percentage of HbA1c | -0.07 (0.08) | -0.87 (0.08)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change from Baseline in Fasting Plasma Glucose collected at Week 16. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline Fasting Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Number analyzed (Participants) | 70 | 77
mg/dL | 8.0 (4.6) | -5.4 (4.4)

3. Secondary Outcome: Change From Baseline in the Areas Under the Curve From 0 to 2 h (AUC0-2h) for Postprandial Plasma Glucose
Description: The change from Baseline in AUC0-2h for Postprandial Plasma Glucose collected at Week 16. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline AUC0-2h for Postprandial Plasma Glucose as a covariate.
Time Frame: 0, 0.5, 1, 2 hours post-dose at Week 0 and Week 16
Population: The full analysis set, consisting of all type 2 diabetic patients, who received at least one dose of study drug and who had at least one efficacy data after randomization.
Measure: Least Squares Mean (Standard Error); unit: mg*hr/dL
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Number analyzed (Participants) | 63 | 74
mg*hr/dL | 9.827 (11.437) | -54.035 (10.552)

4. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose
Description: The change from Baseline in 2-hour Postprandial Plasma Glucose collected at Week 16. Least squares means were derived from an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline 2-hour Postprandial Plasma Glucose as a covariate.
Time Frame: at Week 0 and Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin | Teneli (Teneligliptin) /Teneli + Insulin
Number analyzed (Participants) | 63 | 74
mg/dL | 3.0 (7.6) | -42.9 (7.0)

ADVERSE EVENTS:
Groups:
- Placebo/Teneli (Teneligliptin) + Insulin(Data Through Week 16): Placebo for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained) for an additional 36 weeks (open-label period) in combination with insulin. The adverse events which occured from Week 0 to Week 16 were shown.
- Teneli (Teneligliptin)/Teneli + Insulin(Data Through Week 16): Teneligliptin (20 mg once daily) for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained) for an additional 36 weeks (open-label period) in combination with insulin. The adverse events which occured from Week 0 to Week 16 were shown.
- Placebo/Teneli(Teneligliptin)+Insulin(Data From Week 16 to 52): Placebo for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained) for an additional 36 weeks (open-label period) in combination with insulin. The adverse events which occured from Week 16 to Week 52 were shown.
- Teneli (Teneligliptin) /Teneli + Insulin(Data Through Week 52): Teneligliptin (20 mg once daily) for 16 weeks (double-blind period) followed by teneligliptin (20 mg once daily, titrated to 40 mg if no adequate efficacy is obtained) for an additional 36 weeks (open-label period) in combination with insulin. The adverse events which occured from Week 0 to Week 52 were shown.
Arm/Group | Placebo/Teneli (Teneligliptin) + Insulin(Data Through Week 16) | Teneli (Teneligliptin)/Teneli + Insulin(Data Through Week 16) | Placebo/Teneli(Teneligliptin)+Insulin(Data From Week 16 to 52) | Teneli (Teneligliptin) /Teneli + Insulin(Data Through Week 52)
Serious Adverse Events (participants affected / at risk) | 2/71 | 1/77 | 5/63 | 5/77
Other Adverse Events (participants affected / at risk) | 18/71 | 14/77 | 25/63 | 45/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli (Teneligliptin) + Insulin(Data Through Week 16) (N=71) | Teneli (Teneligliptin)/Teneli + Insulin(Data Through Week 16) (N=77) | Placebo/Teneli(Teneligliptin)+Insulin(Data From Week 16 to 52) (N=63) | Teneli (Teneligliptin) /Teneli + Insulin(Data Through Week 52) (N=77)
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 2
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Teneli (Teneligliptin) + Insulin(Data Through Week 16) (N=71) | Teneli (Teneligliptin)/Teneli + Insulin(Data Through Week 16) (N=77) | Placebo/Teneli(Teneligliptin)+Insulin(Data From Week 16 to 52) (N=63) | Teneli (Teneligliptin) /Teneli + Insulin(Data Through Week 52) (N=77)
Nasopharyngitis (Infections and infestations) | 13 | 6 | 13 | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 9 | 7 | 21
Bronchitis (Infections and infestations) | 1 | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 3 | 4
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 4
Constipation (Gastrointestinal disorders) | 2 | 3 | 3 | 8
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other